CLINICAL TRIAL: NCT02567305
Title: Neutrophil Extracellular Traps and Neonatal (PV4991) & Pediatric Sepsis (PV5063)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4991 & PV5063
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50ul Blood during routine blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Actual Sepsis: For infants below 44 weeks inclusive of corrected age clinical sepsis is defined, according to the Expert Meeting on Neonatal and Pediatric Sepsis (Report on the Expert Meeting on Neonatal and Pediatric Sepsis - 8 June 2010, EMA London). Confirmed sepsis is defined as positive culture for pathogens in a sample from a normally sterile site and at least one laboratory sign or clinical sign (not shown)
  For children above 44 weeks corrected age clinical sepsis is defined according to the Goldstein criteria (Goldstein et al, 2005). Confirmed sepsis: positive culture for pathogens in a sample from a normally sterile site and at least one laboratory sign or clinical sign (not shown)
  Interventions: Other: Markers of NET formation
- Suspected Sepsis: None of the above.
  Interventions: Other: Markers of NET formation

INTERVENTIONS:
Other: Markers of NET formation — i.e. Plasma DNA, Histone, MPO, DNase
  Other Names: Typical biomarkers of NETosis

SUMMARY:
This study is designed to assess the role of neutrophil extracellular traps (NETs) in neonatal and pediatric sepsis as well as to evaluate markers of NETs formation as early predictors of neonatal and pediatric sepsis.

DETAILED DESCRIPTION:
Severe infection resulting in sepsis is recognized as a leading cause of morbidity and mortality worldwide (Stehr and Reinhart, 2013). The incidence of sepsis in developed nations has been increasing while overall mortality is decreasing, but still remains around 30% (Mayr et al., 2014). Moreover, morbidity in survivors is often functionally devastating, and may include neurological impairment, chronic organ dysfunction, increased days admitted to hospital, and high rates of mortality postdischarge (Prescott et al., 2014). Emotional, social, and financial costs to individuals and health care systems are immense (Brun-Buisson et al., 2003).

Neutrophils are the first line of innate immune defense against infectious agents. In addition, neutrophils' ability to eliminate pathogens by phagocytosis and/or degranulation, it has recently been demonstrated that neutrophils can bind to and kill a wide range of microorganisms by forming neutrophil extracellular traps (NETs) (Brinkmann et al., 2004). This novel mechanism consists of the release of web-like structures of DNA decorated with histones and antimicrobial proteins, known as NETs. Microbes are immobilized in these traps, which contain a lethal concentration of antimicrobial agents killing a broad range of microorganisms, including gram-negative and gram-positive bacteria, fungi, viruses, and protozoa (Brinkmann et al., 2004, Fuchs et al., 2010, Camicia et al., 2014).

The role of NETs in pediatric infection is not well understood. We hypnotize that children are capable of forming NETs and that NETosis plays an important role in pediatric sepsis. This study is designed to assess the role of neutrophil extracellular traps (NETs) in neonatal and pediatric sepsis as well as to evaluate markers of NETs formation as early predictors of neonatal and pediatric sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parent or guardian of the patient
2. Chronological age below 90 days (= neonatal branch) or below 18 years (pediatric branch)
3. Suspicion of sepsis infection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children with suspected sepsis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Extracellular Traps | 2 weeks
  Neutrophil Extracellular Traps are measured by serum markers

SECONDARY OUTCOMES:
Sepsis | 2 weeks
  Sepsis is defined according to the Goldstein criteria 2015.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Altona Children's Hospital, Hamburg